CLINICAL TRIAL: NCT03505853
Title: A Drug-Drug Interaction Study to Investigate the Effect of Givosiran on the Pharmacokinetics (PK) of Midazolam, Caffeine, Losartan, Omeprazole, and Dextromethorphan in Patients With Acute Intermittent Porphyria (AIP) Who Are Asymptomatic High Excreters (ASHE)
Brief Title: A Study to Investigate the Interaction Between Givosiran and a 5-probe Drug Cocktail in Patients With Acute Intermittent Porphyria (AIP)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALN-AS1-004
Record Dates: First submitted 2018-04-13; First posted 2018-04-23 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Acute Intermittent Porphyria (AIP); Acute Hepatic Porphyria (AHP); Porphyria, Acute Intermittent; Acute Porphyria
Keywords: RNAi therapeutic; Porphyria; Acute Hepatic Porphyria (AHP); Acute Intermittent Porphyria (AIP)
MeSH Terms: conditions — Porphyria, Acute Intermittent; Coproporphyria, Hereditary; Porphyrias | interventions — givosiran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Givosiran with 5-probe cocktail (Experimental)
  Interventions: Drug: Givosiran; Drug: 5-probe cocktail

INTERVENTIONS:
Drug: Givosiran — single dose of givosiran by subcutaneous (sc) injection
Drug: 5-probe cocktail — includes midazolam, caffeine, losartan, omeprazole, and dextromethorphan

SUMMARY:
The purpose of this study is to evaluate the effect of givosiran on the pharmacokinetics of the 5-probe cocktail of midazolam, caffeine, losartan, omeprazole, and dextromethorphan, and their metabolites, in asymptomatic patients with Acute Intermittent Porphyria.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old
* Weight between 45kg and 110kg, inclusive, if male
* Weight between 45kg and 100 kg, inclusive, if female
* Diagnosis of acute intermittent porphyria (AIP)
* Elevated urine PBG level
* Not be pregnant or breast feeding, and must be willing to use a highly effective method of contraception

Exclusion Criteria:

* Clinically significant abnormal laboratory results
* Experienced an acute porphyria attack within past 12 months
* History of multiple drug allergies, intolerances or sensitivities
* History of recurrent pancreatitis
* Received an experimental drug, within 3 months of dosing
* Donated or lost an excessive amount of blood within 60 days of dosing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Profile of Pharmacokinetics (PK) of Cytochrome P450 (CYP) probe cocktail | Days 1 and 36
  Area under the concentration-time curve (AUC)
Profile of Pharmacokinetics (PK) of Cytochrome P450 (CYP) probe cocktail | Days 1 and 36
  Maximum plasma concentration (Cmax)

SECONDARY OUTCOMES:
Profile of Pharmacokinetics (PK) of Cytochrome P450 (CYP) probe cocktail metabolites | Days 1 and 36
  Area under the concentration-time curve (AUC)
Profile of Pharmacokinetics (PK) of Cytochrome P450 (CYP) probe cocktail metabolites | Days 1 and 36
  Maximum plasma concentration (Cmax)
Profile of Pharmacokinetics (PK) of Cytochrome P450 (CYP) probe cocktail | Days 1 and 36
  Terminal half-life (t1/2)
Profile of Pharmacokinetics (PK) of Cytochrome P450 (CYP) probe cocktail | Days 1 and 36
  Volume of distribution (V/F)
The pharmacodynamic (PD) effect of givosiran on urine levels of delta-aminolevulinic acid (ALA) | Days 1, 8, and 36
The pharmacodynamic (PD) effect of givosiran on urine levels of Porphobilinogen (PBG) in patients with AIP | Days 1, 8, and 36
Safety as evaluated by the proportion of subjects experiencing adverse events (AEs) | Day 1 - Day 92

CONTACTS AND LOCATIONS:
Overall Officials: Nader Najafian, MD, Study Director — Alnylam Pharmaceuticals
Locations (1):
- Clinical Trial Site, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided